CLINICAL TRIAL: NCT03516110
Title: Health Related Quality of Life and Multidimensional Evaluations of a Cohort of Prostate Cancer Subjects Aged ≥ 60 Years Initiating Gonadotropin-Releasing Hormone (GNRH) Agonist Therapy
Brief Title: Health Related Quality of Life and Multidimensional Evaluations of Prostate Cancer Subjects Aged ≥ 60 Years Initiating Gonadotropin-Releasing Hormone (GNRH) Agonist Therapy
Acronym: PRISME
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: A-FR-52014-228
Record Dates: First submitted 2018-03-09; First posted 2018-05-04 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Prostate cancer subjects 60-<70 years
  Interventions: Other: Data collection
- Prostate cancer subjects 70-<75 years
  Interventions: Other: Data collection
- Prostate cancer subjects ≥ 75 years
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Subjects will be treated in accordance with usual medical practice during their participation in this study. No additional assessments or tests will be required.

SUMMARY:
The objective of the study is to compare the evolution over 6 months of Health-Related Quality of Life (HRQOL) among different age groups in subjects with prostate cancer treated with GnRH agonist therapy.

DETAILED DESCRIPTION:
Relevant data collected as part of routine medical care will be captured on an electronic Case Report Form (eCRF). Investigator-subject questionnaires and subject self-questionnaires answers will be collected in a paper booklet. This study is non-interventional, thus if some assessments, are not routinely performed by the investigator, he/she will not complete the corresponding sections in the eCRF.

ELIGIBILITY:
Inclusion Criteria:

* Subject presenting with histologically confirmed prostate cancer
* Subject of 60 years and older
* Subject eligible to start GnRH agonist therapy, either as monotherapy or adjuvant therapy, and for whom one of these treatments was selected voluntarily by the investigator, prior to the start of the study
* Subject giving his written consent to participate in the study
* Subject able to complete questionnaires

Exclusion Criteria:

* Subject simultaneously participating in a clinical trial
* Subject who previously received a hormonal therapy during the last 6 months before inclusion

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate Cancer subjects aged ≥ 60
Sampling Method: Non-Probability Sample
Enrollment: 831 (Actual)
Dates: Start 2018-03-09 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Quality of Life (QOL) as evaluated by Quality of Life Questionnaire-Elderly 14 items (QLQ-ELD-14) | Change from baseline at 6 months
  Evolution overall and in subgroups of age ([60-<70], [70- <75] and ≥ 75 years).

SECONDARY OUTCOMES:
HRQOL Visual Analog Scale (VAS) score | Baseline and 6 months
  Subjects evaluate level of satisfaction with their general health status by indicating a position along a 10 cm-linear analog scale that ranges between 'Not satisfied at all' and 'Totally satisfied'.
Health status scores as evaluated by G8 questionnaire | Baseline and 6 months
Overall condition VAS score | Baseline and 6 months
  Subjects evaluate level of satisfaction with their general health status by indicating a position along a 10 cm-linear analog scale that ranges between 'Not satisfied at all' and 'Totally satisfied'.
Urinary function scores as evaluated by QOL question of the International Prostate Symptom Score (IPSS) | Baseline and 6 months
  Subjects will be asked to indicate the score corresponding to their evaluation of their quality of life related to urinary symptoms in response to the following question 'If you were to live the rest of your life with this way of urinating, would you say you would be:' on a scale from 0 (very satisfied) to 6 (very upset).
Urinary function score VAS | Baseline and 6 months
  Subjects evaluate level of satisfaction with their urinary function by indicating a position along a 10 cm-linear analog scale that ranges between 'Not satisfied at all' and 'Totally satisfied'.
Sexual function scores as evaluated by 3 questions on sexual domain of the Urolife Benign Prostatic Hyperplasia-Quality Of Life 9 (BPH-QoL 9) questionnaire | Baseline and 6 months
Sexual function VAS score | Baseline and 6 months
  Subjects evaluate level of satisfaction with their sexual function by indicating a position along a 10 cm-linear analog scale that ranges between 'Not satisfied at all' and 'Totally satisfied'.
Cognitive status scores as evaluated by Mini Mental State (MMS) | Baseline and 6 months
Memory VAS score | Baseline and 6 months
  Subjects evaluate level of satisfaction with memory (your capacity to remind events or persons you meet) by indicating a position along a 10 cm-linear analog scale that ranges between 'Not satisfied at all' and 'Totally satisfied'.
Mood scores as evaluated by mini Geriatric Depression Scale (GDS) questionnaire | Baseline and 6 months
  Subjects will be asked four questions and their responses 'Yes' or 'No' will be scored from 0 to 1.
Mood VAS score | Baseline and 6 months
  Subjects evaluate level of satisfaction with mood (your feeling of happiness, confidence and serenity) by indicating a position along a 10 cm-linear analog scale that ranges between 'Not satisfied at all' and 'Totally satisfied'.
Motricity scores as evaluated by G8 questionnaire specific domain (3rd item) | Baseline and 6 months
  Mobility will be scored as follows 'Bed or chair bound' = 0, 'Able to get out of bed/chair but does not go out' = 1, 'Goes out' = 2
VAS motricity score | Baseline and 6 months
  Subjects evaluate level of satisfaction with motricity (your ability to move by yourself in your home or outside) by indicating a position along a 10 cm-linear analog scale that ranges between 'Not satisfied at all' and 'Totally satisfied'
Autonomy question | Baseline and 6 months
  Subjects respond either 'yes' or 'no' to the following autonomy question 'Is the patient living independently at home?'
Autonomy VAS score | Baseline and 6 months
  Subjects evaluate level of satisfaction with autonomy (your ability to manage your life alone at home or outside) by indicating a position along a 10 cm-linear analog scale that ranges between 'Not satisfied at all' and 'Totally satisfied'.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Ipsen Central Contact, Paris, France